CLINICAL TRIAL: NCT05569707
Title: MR Lymphography and Magnetic Sentinel Lymph Node Biopsy in Melanoma Patients Measured With DiffMag
Brief Title: MR Lymphography and Magnetic Sentinel Lymph Node Biopsy in Melanoma Patients
Acronym: MelaDiff
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Twente (Other)
Responsible Party: Principal Investigator, Anke Christenhusz, PhD student / coordinating investigator, University of Twente
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL79537.100.21
Record Dates: First submitted 2022-09-17; First posted 2022-10-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Melanoma (Skin)
Keywords: Magnetic sentinel lymph node biopsy (SLNB); Lymph node detection; Lymph node staging; MR lymphography; Super paramagnetic iron-oxide (SPIO) nanoparticles
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MelaDiff (Other): Patients with melanoma of the extremities included in the protocol. Preoperative, patients will receive two MRI-scans and a magnetic tracer injection at the primary tumor site. During surgery, SLNs will be detected using two types of magnetometers (SentiMag® & DiffMag) in combination with Magtrace®, in addition to the standard procedure.
  Interventions: Device: Magnetic sentinel lymph node biopsy by use of Magtrace®, in combination with SentiMag® and DiffMag

INTERVENTIONS:
Device: Magnetic sentinel lymph node biopsy by use of Magtrace®, in combination with SentiMag® and DiffMag — In addition to the standard procedure, SLNs will be detected using two types of magnetometers (SentiMag® & DiffMag) in combination with SPIO particles (Magtrace®).

SUMMARY:
The sentinel lymph nodes (SLNs) are the first lymph nodes (LNs) to drain the tumor site and therefore the first LNs to bare metastases. Hence the importance to investigate these LNs for the best treatment strategy. Current-standard-of-care for melanoma patients with a melanoma stage of pT1b or higher, involve a surgical procedure, referred to as SLN biopsy (SLNB). The SLNB procedure involves a combined detection procedure using a radio-active tracer and blue dye followed by surgical dissection and evaluation of the LNs at the histopathology department. Due to the use of radioisotopes, this procedure suffers from several disadvantages such as limited availability, strict rules and regulations, degradation time in patient and radioactive load for user and patient.

To overcome the limitations of a radioactive tracer, a magnetic SLNB was developed which is facilitated by super paramagnetic iron-oxide (SPIO) nanoparticles. This potentially offers numerous benefits making surgery planning more flexible: no exposure to radiation, easy accessibility of the tracer, long shelf life and long half time in the patient. However, the currently available magnetometer for intraoperative detection of SPIO-enhanced LNs is hampered by a relatively low detection depth, biological noise, and effects of surgical equipment. Therefore, surgeons need to switch to plastic or carbon equipment and the system needs to be balanced prior to each measurement, which increases the surgery time.

A new and effective way to localize SPIOs is differential magnetometry (DiffMag). This patented detection principle, developed by MD&I group at University of Twente (UT), utilizes the nonlinear magnetic response of nanoparticles. An additional advantage of SPIOs is their visibility on MRI, which could provide mapping the SLNs preoperatively. Especially in patients with melanomas on the abdomen or back this would be very useful to see which lymph node stations are connected to the melanoma. In addition, studies have shown that SPIOs are absorbed into lymph nodes in different ways, depending on the presence of metastases. SPIO-enhanced MR lymphography could therefore provide an opportunity for a non-invasive preoperative assessment of nodal status.

In this pilot study the investigators want to evaluate the clinical use of the DiffMag handheld probe. Moreover, the investigators want to map the lymph nodes (metastases) preoperatively using MR lymphography.

ELIGIBILITY:
Inclusion Criteria:

* Patients with melanoma of the upper or lower extremities scheduled for SLNB;
* Willing to & able to write informed consent from the subject prior to participation;
* Willing to & capable of following study procedures;
* Is older than 18 years;
* Speaks and understand the Dutch language

Exclusion Criteria:

* Intolerance / hypersensitivity to iron or dextran compounds
* Pregnant or lactating patients;
* Patients having a pacemaker.
* Patients non eligible for MRI investigation (pacemakers or other implantable devices in the chest wall and/or lower body, claustrophobic, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
True positive/False negative rate for a magnetic SLN detection measured by DiffMag system compared to radioactive detection. | through study completion, an average of 1 year
  Determining the feasibility of SLN detection/localization in melanoma patients using a magnetic tracer (Magtrace®) and hand-held magnetometer DiffMag.
True positive/False negative rate for a magnetic SLN detection measured by Sentimag system compared to radioactive detection. | through study completion, an average of 1 year
  Determining the feasibility of SLN detection/localization in melanoma patients using a magnetic tracer (Magtrace®) and hand-held magnetometer Sentimag.

SECONDARY OUTCOMES:
True positive/False negative rate for metastatic SLN using ex vivo MRI | through study completion, an average of 1 year
  Determining the feasibility of LN mapping with preoperative SPIO-enhanced MR lymphography and examining the use of SPIO-enhanced MR lymphography for LN staging.
True positive/False negative rate for metastatic SLN using in vivo MRI | through study completion, an average of 1 year
  Determining the feasibility of LN mapping with preoperative SPIO-enhanced MR lymphography and examining the use of SPIO-enhanced MR lymphography for LN staging.

CONTACTS AND LOCATIONS:
Overall Officials: Lejla Alic, PhD, Study Chair — University of Twente; Anneriet Dassen, PhD, Principal Investigator — Medisch Spectrum Twente Enschede
Locations (2):
- Netherlands (2):
  - Medisch Spectrum Twente, Enschede
  - Ziekenhuisgroep Twente (ZGT), Hengelo

IPD SHARING:
Plan to Share IPD: No